CLINICAL TRIAL: NCT04278599
Title: Comparative Evaluation of Effect of Oral Zinc Supplementation and Placebo as an Adjuvant to Topical Corticosteroid Therapy in Oral Lichen Planus Patients
Brief Title: Effect of Oral Zinc Supplementation as an Adjuvant to Topical Corticosteroid in Oral Lichen Planus Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: shagun257
Record Dates: First submitted 2020-02-18; First posted 2020-02-20 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Oral Lichen Planus
MeSH Terms: conditions — Lichen Planus, Oral | interventions — Zinc Acetate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental): The patients will be administered Zinc Acetate tablets (equivalent to 30 mg of elemental zinc/day) for 6 weeks from the baseline. Topical corticosteroid paste will be prescribed according to the intensity of the lesion.
  Interventions: Drug: Oral Zinc supplementation
- Control group (Placebo Comparator): The patients will be administered Placebo tablets for 6 weeks from the baseline. Topical corticosteroid paste will be prescribed according to the intensity of the lesion.
  Interventions: Drug: Oral placebo supplementation

INTERVENTIONS:
Drug: Oral Zinc supplementation — In the test group, the patients will be administered Zinc Acetate tablets (equivalent to 30 mg of elemental zinc/day) for 6 weeks from the baseline. They will also be will be administered, topical corticosteroid paste- Triamcinolone acetonide- 0.1%, to be applied thrice a day till the lesions disappeared and the dosage will be tapered accordingly.The patients will be instructed to take the tablets and apply the paste after meals.The patients will be kept on a monthly follow-up for 3 months.
  Other Names: Zinc Acetate
  Arms: Test group
Drug: Oral placebo supplementation — In the control group, the patients will be administered Placebo tablets for 6 weeks from the baseline. They will also be administered, topical corticosteroid paste- Triamcinolone acetonide- 0.1%, to be applied thrice a day till the lesions disappeared and the dosage will be tapered accordingly.The patients will be instructed to take the tablets and apply the paste after meals.The patients will be kept on a monthly follow-up for 3 months.
  Other Names: Placebo
  Arms: Control group

SUMMARY:
Lichen planus is an auto-immune, chronic inflammatory disease that affects mucosal and cutaneous tissue. Erosive and atrophic oral lichen planus (OLP) are difficult to manage because patients present with symptoms ranging from episodic pain to severe discomfort and they have the highest malignant transformation rate (MTR) amongst all the forms of OLP. Zinc is associated with regeneration of epithelium, wound healing and mediating T-lymphocyte function; all of which can lead to healing and re-epithelisation in the lesions of erosive OLP. Besides this, it also has anti-oxidant and anti-inflammatory properties, which lead to decrease in apoptosis and transformation into a malignant state.

This study intends to evaluate the effect of oral zinc supplements as an adjuvant to the topical corticosteroid therapy in the treatment of OLP.

DETAILED DESCRIPTION:
Lichen planus is a chronic muco-cutaneous disorder of the stratified squamous epithelium that affects the oral and genital mucous membrane, skin, hair, nails and scalp.OLP is the mucosal counterpart of cutaneous lichen planus.The disease was first described by Erasmus Wilson in 1866. The prevelance of disease in the Indian sub-continent is about 2.6%,with the mean age being 30-60 years and with a female predilection. The cutaneous form is more persistent and resistant to treatment while OLP is more frequent in occurrence.

OLP is a potentially pre-malignant oral epithelial lesion. It is a T-cell mediated auto-immune disease in which the auto-cytotoxic CD8 + T cells trigger the apoptosis of the basal cells of oral epithelium.OLP is an idiopathic disease, although there are certain precipitating factors like HLA-A3, anxiety & stress, diabetes and hypertension.

OLP occurs bilaterally, the most common sites being buccal mucosa, tongue, lips, gingiva, floor of mouth and palate. Wickham's striae are a pathogonomic feature. It has six clinical presentations- Reticular, Erosive, Atrophic, Plaque-like, Papular and Bullous.The reticular form is most common but its asymptomatic, while the erosive form is most severe with symptoms ranging from mild burning to severe pain. The range of MTR for OLP is about 0-5%, with the highest rate for erosive and atrophic types.Erosive OLP lesions arise as a complication of the atrophic process after trauma or ulceration. Appear as a central area of erosion with yellowish fibrinous exudate surrounded by erythema, with Wickham's striae in the periphery. Atrophic OLP lesions appear bright red due to loss of epithelium.

A review study done on the recent concepts in the treatment of OLP concluded that corticosteroids (mostly topical, rarely systemic) continue to be the mainstay of management of OLP. However, there are some other drugs which have a significant contribution such as- Calcineurin inhibitors (cyclosporine, tacrolimus, pimecrolimus), Retinoids, Dapsone, Hydroxychloroquine, Mycophenolate mofetil and Enoxaprin. The non-pharmacological treatment modalities include PUVA therapy, photodynamic therapy and laser therapy.

A recently conducted study found out that serum zinc levels were significantly decreased in patients with erosive OLP in comparison with patients of non-erosive OLP, which may be responsible for disintegration of epithelium in erosive OLP lesions.

The association of OLP and zinc lies in the fact that zinc is associated with the regeneration of epithelium, enhancement of enzyme activity, contributes to protein structure, helps in wound healing as well as inhibition and stimulation of lymphocyte reaction.The deficiency of zinc also leads to compromised T-cell mediated immune defence.Zinc also has anti-oxidant and anti-inflammatory properties, which can decrease apoptosis and transformation to a malignant state.

Thus, the present study intends to evaluate the role of oral zinc supplementation as an adjuvant to topical corticosteroid therapy on the treatment of oral lichen planus.

ELIGIBILITY:
Inclusion Criteria:

1. Clinically and histopathologically proven cases of erosive and atrophic OLP.
2. Patients who are willing to participate in the study.

Exclusion Criteria:

1. Patients with reticular form of OLP and OLP with muco-cutaneous involvement.
2. Patients consuming drugs for the treatment of OLP in the past 6 months.
3. Suspected lichenoid reaction associated with drugs and restorations.
4. Patients whose histopathological findings indicate moderate to severe dysplasia.
5. Patients with acquired and congenital immuno-deficiency disorders like AIDS, chemotherapy, addiction to injectable opioids like hemophilia and blood dialysis. These patients are excluded because of difficulty in their biopsy procedure, control of infection, possible interaction with clinical findings of OLP, and their potential doubtful cooperation.
6. Patients with systemic diseases involving the gastro-intestinal tract.
7. Known cases of Acrodermatitis enteropathica where difficulty in zinc absorption persists.
8. Presence of factors that can alter the absorption of zinc like consumption of calcium tablets, iron supplements and high protein diet.
9. Pregnancy and lactation phase
10. Alcoholic patients, since alcoholism results in intracellular zinc deficiency.
11. Recorded allergy to zinc and/or corticosteroids.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2020-01-15 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Assessment of changes in size of the lesion | Baseline, 6 weeks and 3 months.
  Thongprasom score (TS) will be used to assess changes in the size of the lesion. Digital Vernier callipers will be used to measure the largest dimension of ulcers at baseline and at each follow-up visit.
Assessment of changes in pain and burning sensation of the lesion. | Baseline, 6 weeks and 3 months
  Visual Analogue Scale (VAS) will be used to assess changes in pain and burning sensation of the lesion.
Assessment of changes in changes in erythema and ulceration. | Baseline, 6 weeks and 3 months
  Modified Oral Mucositis Index (MOMI)- will be used to assess changes in erythema and ulceration.
Assessment of quality of life of the patient. | Baseline, 6 weeks and 3 months
  Oral Health Impact Profile -14 index (OHIP-14) will be used to assess the quality of life of the patient.

SECONDARY OUTCOMES:
Number of episodes of new lesions in the follow-up period. | Baseline, 6 weeks and 3 months
  The frequency of episodes of new lesions in the follow-up period will be assessed by visual examination
Adverse effects of oral zinc supplementation. | Baseline, 6 weeks and 3 months
  The will adverse effects of oral zinc supplementation.be assessed by interviewing the patients
Requirement for additional systemic steroid therapy. | Baseline, 6 weeks and 3 months
  The requirement for additional systemic steroid therapy will be decided by the presence of non-healing ulcers with persistent VAS scores

CONTACTS AND LOCATIONS:
Overall Officials: Shagun Solanki, Principal Investigator — Post Graduate Institute of Dental Sciences, Rohtak
Locations (1):
- Post Graduate Institute of Dental Sciences, Rohtak, Haryana, India